CLINICAL TRIAL: NCT07156656
Title: Assessment of the Efficacy of Sivelestat Sodium Treatment in Post-operative Organ Dysfunction in Patients With Acute Type A Aortic Dissection (STOP): a Multicenter, Double-blind RCT
Brief Title: Sivelestat Treatment for Postoperative Organ Protection in Type A Aortic Dissection
Acronym: STOP
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: The First Affiliated Hospital of Anhui Medical University (Other); Fujian Provincial Hospital (Other); The University of Hong Kong-Shenzhen Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Guangdong Provincial People's Hospital (Other); Changhai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B2025-349R
Record Dates: First submitted 2025-08-20; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Type A Aortic Dissection; Organ Failure, Multiple
Keywords: Type A Aortic Dissection; SOFA; Sivelestat Sodium; Multiple Organ Failure
MeSH Terms: conditions — Multiple Organ Failure

STUDY DESIGN:
Intervention Model Description: a Multicenter, Double-blind RCT
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sivelestat group (Experimental): Drug: Sivelestat Sodium. Procedure: Conventional Treatment
  Interventions: Procedure: Conventional treatment; Drug: Sivelestat sodium
- Control group (Placebo Comparator): Drug: Placebo. Procedure: Conventional Treatment
  Interventions: Procedure: Conventional treatment; Drug: Placebo

INTERVENTIONS:
Procedure: Conventional treatment — Beside the using of Sivelestat Sodium or placebo, all postoperative care will adhere to each center's standard protocols for type A aortic dissection.
Drug: Sivelestat sodium — The daily dose (4.8 mg/kg) is diluted in 48 mL of 0.9 % saline and administered as a continuous intravenous infusion over 24 hours at 2 mL/h (equivalent to 0.2 mg/kg/h) for 72 consecutive hours.
  Other Names: Siv
  Arms: Sivelestat group
Drug: Placebo — An equal volume of placebo-containing only the excipients of sivelestat sodium and diluted to 48 mL with 0.9 % saline-will be infused at 2 mL/h for 72 consecutive hours.
  Arms: Control group

SUMMARY:
The goal of this multicenter, double-blind, randomized controlled trial is to learn if sivelestat sodium (Siv) can protect the organ function in patients suffered operation for acute type A aortic dissection. The main questions it aims to answer are:

* Can the 3-day-treatment of Siv enlarge the Day-0-to-Day-5 drop in the organ-health score (SOFA score)?
* Can this treatment significantly shrink the area under the SOFA curve from first dose to Day 5?
* Can this treatment significantly improve the end of patients in 28 days (clinical outcomes)? Researchers will compare drug Siv to a placebo (a look-alike substance that contains no drug) to see if drug Siv works.

Participants will:

* Take drug Siv or the placebo through vein continuously for 72 hours
* Receiving regular intensive care in ICU after the operation

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years inclusive.
2. Written informed consent obtained before participation.
3. Confirmed acute Stanford type A aortic dissection scheduled for surgical repair.

Exclusion Criteria:

1. Life expectancy ≤ 48 hours.
2. Pregnant or lactation.
3. Severe pre-operative liver dysfunction: Child-Turcotte-Pugh score 10-15.
4. Severe pre-operative renal dysfunction: acute or chronic kidney injury meeting criteria for renal-replacement therapy.
5. Confirmed COPD or asthma.
6. Immunosuppression: long-term or > 2 weeks continuous systemic corticosteroids.
7. Concomitant or anticipated use of immunomodulators (Xue-Bi-Jing injection, thymosin, IVIG).
8. Medical or psychological condition that would interfere with study participation, assessment, or outcomes.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
ΔSOFA5 | from the entry of ICU(baseline, post-operatively) to the fifth day in ICU(the fifth day after the first dose)
  ΔSOFA5 is defined as the decrease level of SOFA(Sequential Organ Failure Assessment) score from baseline to the fifth day. SOFA score ranges from 0~24, the higher the score, the poorer the functionality of multiple organs.

SECONDARY OUTCOMES:
AUC - SOFA | from the entry of ICU(baseline, post-operatively) to the fifth day in ICU(the fifth day after the first dose)
  Area under the SOFA-time curve
Clinical Outcomes - Incidence of tracheotomy | from the entry of ICU(baseline, post-operatively) to the 28th day after surgery
  Incidence of tracheotomy
Clinical Outcomes - Re-intubation rate | from the entry of ICU(baseline, post-operatively) to the 28th day after surgery
  Re-intubation rate
Clinical Outcomes - Gastrointestinal bleeding （count, rate） | from the entry of ICU(baseline, post-operatively) to the 28th day after surgery
  Gastrointestinal bleeding （count, rate）
Clinical Outcomes - Infection | from the entry of ICU(baseline, post-operatively) to the 28th day after surgery
  Infection: Serious infections such as bloodstream infections, sepsis, ventilator-associated pneumonia
Clinical Outcomes - In-hospital mortality | from the entry of ICU(baseline, post-operatively) to the 28th day after surgery
  In-hospital mortality
Clinical Outcomes - ICU length of stay (days) | from the entry of ICU(baseline, post-operatively) to the 28th day after surgery
  ICU length of stay (days)
Clinical Outcomes - Total hospital length of stay (days) | from the entry of ICU(baseline, post-operatively) to the 28th day after surgery
  Total hospital length of stay (days)
Clinical Outcomes - Ventilator-free days at day 28 (days) | from the entry of ICU(baseline, post-operatively) to the 28th day after surgery
  Mechanical ventilation includes: invasive mechanical ventilation and non-invasive mechanical ventilation
Clinical Outcomes - Invasive ventilatory support duration at day 28 (days) | from the entry of ICU(baseline, post-operatively) to the 28th day after surgery
  Invasive ventilatory support: invasive mechanical ventilation
Clinical Outcomes - Respiratory-support-free time at day 28 (days) | from the entry of ICU(baseline, post-operatively) to the 28th day after surgery
  Respiratory support includes: invasive mechanical ventilation, non-invasive mechanical ventilation, and high-flow oxygen
Clinical Outcomes - Organ-support-free days at day 28(days) | from the entry of ICU(baseline, post-operatively) to the 28th day after surgery
  days free of mechanical ventilation, vasopressors, and renal-replacement therapy
Clinical Outcomes - Central nervous system complications during ICU stay | from the entry of ICU(baseline, post-operatively) to the 28th day after surgery
  Central nervous system complications during ICU stay: cerebral infarction, intracranial hemorrhage, hypoxic-ischemic encephalopathy
Clinical Outcomes - Delirium incidence during ICU stay | from the entry of ICU(baseline, post-operatively) to the 28th day after surgery
  Delirium incidence during ICU stay
Clinical Outcomes - Incidence of acute kidney injury (AKI) | from the entry of ICU(baseline, post-operatively) to the 28th day after surgery
  Incidence of acute kidney injury (AKI)
Laboratory Test Results - Arterial blood gas: pH | from the entry of ICU(baseline, post-operatively) to the fifth day in ICU(the fifth day after the start of treatment)
  pH result from arterial blood gas
Laboratory Test Results - Arterial blood gas: PaO₂/FiO₂ | from the entry of ICU(baseline, post-operatively) to the fifth day in ICU(the fifth day after the start of treatment)
  PaO₂/FiO₂ result from arterial blood gas
Laboratory Test Results - Arterial blood gas: SpO₂/FiO₂ | from the entry of ICU(baseline, post-operatively) to the fifth day in ICU(the fifth day after the start of treatment)
  SpO₂/FiO₂ result from arterial blood gas
Laboratory Test Results - Arterial blood gas: PaO₂ | from the entry of ICU(baseline, post-operatively) to the fifth day in ICU(the fifth day after the start of treatment)
  PaO₂ result from arterial blood gas
Laboratory Test Results - Arterial blood gas: PaCO₂ | from the entry of ICU(baseline, post-operatively) to the fifth day in ICU(the fifth day after the start of treatment)
  PaCO₂ result from arterial blood gas
Laboratory Test Results - Arterial blood gas: SpO₂ | from the entry of ICU(baseline, post-operatively) to the fifth day in ICU(the fifth day after the start of treatment)
  SpO₂ result from arterial blood gas
Laboratory Test Results - Arterial blood gas: lactate | from the entry of ICU(baseline, post-operatively) to the fifth day in ICU(the fifth day after the start of treatment)
  lactate result from arterial blood gas
Laboratory Test Results - Liver & kidney function: AST | from the entry of ICU(baseline, post-operatively) to the fifth day in ICU(the fifth day after the start of treatment)
  AST from Liver & kidney function
Laboratory Test Results - Liver & kidney function: ALT | from the entry of ICU(baseline, post-operatively) to the fifth day in ICU(the fifth day after the start of treatment)
  ALT from Liver & kidney function
Laboratory Test Results - Liver & kidney function: ALP | from the entry of ICU(baseline, post-operatively) to the fifth day in ICU(the fifth day after the start of treatment)
  ALP from Liver & kidney function
Laboratory Test Results - Liver & kidney function: GGT | from the entry of ICU(baseline, post-operatively) to the fifth day in ICU(the fifth day after the start of treatment)
  GGT from Liver & kidney function
Laboratory Test Results - Liver & kidney function: TBil | from the entry of ICU(baseline, post-operatively) to the fifth day in ICU(the fifth day after the start of treatment)
  TBil from Liver & kidney function
Laboratory Test Results - Liver & kidney function: DBIL | from the entry of ICU(baseline, post-operatively) to the fifth day in ICU(the fifth day after the start of treatment)
  DBIL from Liver & kidney function
Laboratory Test Results - Liver & kidney function: ALB | from the entry of ICU(baseline, post-operatively) to the fifth day in ICU(the fifth day after the start of treatment)
  ALB from Liver & kidney function
Laboratory Test Results - Liver & kidney function: Scr | from the entry of ICU(baseline, post-operatively) to the fifth day in ICU(the fifth day after the start of treatment)
  Scr from Liver & kidney function
Laboratory Test Results - Liver & kidney function: BUN | from the entry of ICU(baseline, post-operatively) to the fifth day in ICU(the fifth day after the start of treatment)
  BUN from Liver & kidney function
Laboratory Test Results - Liver & kidney function: eGFR | from the entry of ICU(baseline, post-operatively) to the fifth day in ICU(the fifth day after the start of treatment)
  eGFR from Liver & kidney function
Laboratory Test Results - Liver & kidney function: NGAL | from the entry of ICU(baseline, post-operatively) to the fifth day in ICU(the fifth day after the start of treatment)
  NGAL from Liver & kidney function
Laboratory Test Results - Myocardial injury: CK-MB | from the entry of ICU(baseline, post-operatively) to the fifth day in ICU(the fifth day after the start of treatment)
  CK-MB from Myocardial injury
Laboratory Test Results - Myocardial injury: LDH | from the entry of ICU(baseline, post-operatively) to the fifth day in ICU(the fifth day after the start of treatment)
  LDH from Myocardial injury
Laboratory Test Results - Myocardial injury: cTnI or cTnT | from the entry of ICU(baseline, post-operatively) to the fifth day in ICU(the fifth day after the start of treatment)
  cTnI or cTnT from Myocardial injury
Laboratory Test Results - Myocardial injury: BNP or NT-proBNP | from the entry of ICU(baseline, post-operatively) to the fifth day in ICU(the fifth day after the start of treatment)
  BNP or NT-proBNP from Myocardial injury
Laboratory Test Results - Brain injury: NSE | from the entry of ICU(baseline, post-operatively) to the fifth day in ICU(the fifth day after the start of treatment)
  NSE result from blood test, Brain injury part
Laboratory Test Results - Inflammation: CRP | from the entry of ICU(baseline, post-operatively) to the fifth day in ICU(the fifth day after the start of treatment)
  CRP result from Inflammation test
Laboratory Test Results - Inflammation: PCT | from the entry of ICU(baseline, post-operatively) to the fifth day in ICU(the fifth day after the start of treatment)
  PCT result from Inflammation test
Laboratory Test Results - Inflammation: IL-6 | from the entry of ICU(baseline, post-operatively) to the fifth day in ICU(the fifth day after the start of treatment)
  IL-6 result from Inflammation test8
Laboratory Test Results - Inflammation: IL-8 | from the entry of ICU(baseline, post-operatively) to the fifth day in ICU(the fifth day after the start of treatment)
  IL-8 result from Inflammation test
Laboratory Test Results - Inflammation: IL-10 | from the entry of ICU(baseline, post-operatively) to the fifth day in ICU(the fifth day after the start of treatment)
  IL-10 result from Inflammation test
Laboratory Test Results - Inflammation: TNF-α | from the entry of ICU(baseline, post-operatively) to the fifth day in ICU(the fifth day after the start of treatment)
  TNF-α result from Inflammation test

OTHER OUTCOMES:
Plasma neutrophil elastase levels (exploratory outcome) | from the entry of ICU(baseline, post-operatively) to the fifth day in ICU(the fifth day after the first dose)
  Plasma concentration of neutrophil elastase at 1day, 3day and 5day after the first dose in 40 participants enrolled at the main center (20 per arm).

CONTACTS AND LOCATIONS:
Overall Officials: Zhe Luo, Study Chair — Fudan University
Locations (6):
- China (6):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Fujian Provincial Hospital, Fuzhou, Fujian
  - Guangdong Provincial People's Hospital (Guangdong Academy of Medical Sciences) (Guangdong Provincial People's Hospital Affiliated to Southern Medical University), Guangzhou, Guangdong
  - The University of Hong Kong - Shenzhen Hospital, Shenzhen, Guangdong
  - The First Affiliated Hospital of Xi'an Jiao Tong University, Xi'an, Shaanxi
  - Changhai Hospital of Shanghai, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No